CLINICAL TRIAL: NCT06272552
Title: Implementing PROMs and PREMs in Routine Clinical Care: Assessment of Requirements and Impact.
Acronym: PROMs & PREMs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PI21-00026; 2021/10182/I (Other: CEIm Parc de Salut Mar)
Record Dates: First submitted 2024-02-12; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: PROMs; PREMs; Implementation Research; Impact Evaluation
Keywords: PRMs Implementation; Implementation Research; Implementation evaluation; PROMs; PREMs; Impact evaluation; RCT; Health Services Research
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PROMs and PREMs (Experimental)
  Interventions: Other: PROMs and PREMs
- PREMs (Active Comparator)
  Interventions: Other: PREMs
- Control (Active Comparator)
  Interventions: Other: Control
- Healthcare professionals (Other)
  Interventions: Other: Healthcare professionals

INTERVENTIONS:
Other: PROMs and PREMs — Participants are administered PROMs and PREMs at a given timeline adequate to each participant conditions for a duration of 2 years. The administration of PROMs is done by email using the REDCap platform. The research team and health care professionals have access to their patient's results to aid in the patients clinical care.
  Participants are administered a PREM once a year for two years. Only health care administrators, department heads and researchers will have access to the PREMs data, and this data will always be aggregated data to avoid identification of the patients. The administration of the PREM is done by email using the REDCap platform.
  At recruitment and once a year, participants answer an evaluation questionnaire to measure the impact of completing PROMs and PREMs. This questionnaire is completed during a clinic visit.
  Arms: PROMs and PREMs
Other: PREMs — Participants are administered a PREM once a year for two years. Only health care administrators, department heads and researchers will have access to the PREMs data, and this data will always be aggregated data to avoid identification of the patients. The administration of the PREM is done by email using the REDCap platform.
  At recruitment and once a year, participants answer an evaluation questionnaire to measure the impact of completing PROMs and PREMs. This questionnaire is completed during a clinic visit.
  Arms: PREMs
Other: Control — At recruitment and once a year, participants answer an evaluation questionnaire to measure the impact of completing PROMs and PREMs. This questionnaire is completed during a clinic visit.
  Arms: Control
Other: Healthcare professionals — Healthcare professionals participating in the study answer an evaluation questionnaire before the implementation starts at their service and two years later to measure their perceptions about the implementation.
  Arms: Healthcare professionals

SUMMARY:
There has been increasing interest in the use of patient-reported outcomes and experience measures (PROMs and PREMs) in clinical practice; yet few empirical studies have been conducted to evaluate the usefulness of such implementation.

Objective: To evaluate the efficacy of the implementation of PROMs and PREMs in routine clinical care for improving health outcomes and satisfaction with health management.

Design: Randomized control trial. Setting: In and outpatient departments of a public hospital in Spain.

Participants: 1,440 adult patients managed for breast cancer, prostate cancer, chronic kidney disease, or bariatric surgery.

Intervention: Patients will monthly complete, through an App from their smartphones, PROMs and PREMs (arm A, n=480), or only PREMs (arm B, n=480). Responses to PROMs will be transformed into a graphic summary, accessible for physicians and patients at the follow-up visits of the project (9 and 18 months after recruitment).

Main outcome measures: Comparison of change among arms on the assessment variables - such as health-related quality of life (EQ-5D-5L), satisfaction with care, or patient-professionals communication. These constructs will be measured at recruitment and at follow up visits for all patients, regardless of their arm allocation (arm C would only be administered these questionnaires, without intervention, n=480).

Expected results: Incorporating PROMs and PREMs in routine clinical care may improve patients' and health professionals' experiences on health care, as well as improve patients' health.

ELIGIBILITY:
Inclusion Criteria:

* Being an active patient of the nephrology service, prostate cancer service, breast cancer service, or bariatric surgery service
* In possession of an email account and having basic knowledge of how to manage emails
* In possession of a smartphone, computer, or tablet with access to the Internet
* Fluent and able to read in Spanish

Exclusion Criteria:

- Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation quesionnaire (PRMIAT) of the implementation to be completed by all patients and healthcare professionals | At recruitment and at 1 year intervals
  The PRMIAT measures the perceptions of the patients and healthcare professionals about the implementation of PROMs and PREMs in routine clinical care
Health-related quality of life | At recruitment and at 1 year intervals
  Measured with the EQ-5D-5L in all patients that participate.

CONTACTS AND LOCATIONS:
Overall Officials: Olatz Garin, PhD, Principal Investigator — Hospital del Mar Research Institute
Locations (1):
- Hospital del Mar Reseach Institute, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon request to outside institutions after data from all individual patients has been anonimized and once the study has finalized and main results have been published.